CLINICAL TRIAL: NCT00267280
Title: A Phase 3, Open-Label, Multisite, Randomized, Parallel Group Study of the Efficacy and Safety of Fixed Combination Torcetrapib/Atorvastatin Administered Once Daily (QD) Compared to Simvastatin for 6 Weeks in Subjects With Hypercholesterolemia (A5091031)
Brief Title: A Clinical Trial Comparing Torcetrapib/Atorvastatin To Simvastatin In Subjects With High Cholesterol (A5091031).
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A5091031
Record Dates: First submitted 2005-12-19; First posted 2005-12-20 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Hyperlipidemia; Dyslipidemia; Hypercholesterolemia
MeSH Terms: conditions — Hyperlipidemias; Dyslipidemias; Hypercholesterolemia | interventions — torcetrapib; Atorvastatin; Simvastatin

INTERVENTIONS:
Drug: torcetrapib/atorvastatin
Drug: simvastatin

SUMMARY:
The Torcetrapib project was terminated on December 2, 2006 due to safety findings.

Cholesterol levels will be measured over six weeks in subjects being treated with two different kinds of cholesterol medications to see how the different treatments compare to one another.

DETAILED DESCRIPTION:
For additional information please call: 1-800-718-1021

ELIGIBILITY:
Inclusion Criteria:

* eligible for statin treatment for LDL cholesterol by NCEP guidelines

Exclusion Criteria:

* Women who are pregnant or lactating, or planning to become pregnant.
* Subjects taking any drugs known to be associated with an increased risk of myositis in combination with HMG-CoA reductase inhibitors.
* Subjects with significant liver or kidney disease or significant heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640
Dates: Start 2006-01; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Percent change in LDL-C and HDL-C from baseline, after six weeks of treatment.

SECONDARY OUTCOMES:
Changes in other lipid parameters and other biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (51):
- United States (51):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Mesa, Arizona
  - Pfizer Investigational Site, Alhambra, California
  - Pfizer Investigational Site, Inglewood, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Santa Ana, California
  - Pfizer Investigational Site, Wilmington, Delaware
  - Pfizer Investigational Site, Fort Lauderdale, Florida
  - Pfizer Investigational Site, Hollywood, Florida
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Merritt Island, Florida
  - Pfizer Investigational Site, Pensacola, Florida
  - Pfizer Investigational Site, Vero Beach, Florida
  - Pfizer Investigational Site, Winter Park, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Conyers, Georgia
  - Pfizer Investigational Site, Woodstock, Georgia
  - Pfizer Investigational Site, Hinsdale, Illinois
  - Pfizer Investigational Site, La Grange, Illinois
  - Pfizer Investigational Site, Park Ridge, Illinois
  - Pfizer Investigational Site, Springfield, Illinois
  - Pfizer Investigational Site, Kansas City, Kansas
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Bethesda, Maryland
  - Pfizer Investigational Site, Elkton, Maryland
  - Pfizer Investigational Site, Flint, Michigan
  - Pfizer Investigational Site, Springfield, Missouri
  - Pfizer Investigational Site, Lawrenceville, New Jersey
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Seaford, New York
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Mansfield, Ohio
  - Pfizer Investigational Site, Hillsboro, Oregon
  - Pfizer Investigational Site, Beaver, Pennsylvania
  - Pfizer Investigational Site, Flourtown, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Yardley, Pennsylvania
  - Pfizer Investigational Site, Greenville, South Carolina
  - Pfizer Investigational Site, Collierville, Tennessee
  - Pfizer Investigational Site, Kingsport, Tennessee
  - Pfizer Investigational Site, Knoxville, Tennessee
  - Pfizer Investigational Site, North Richland Hills, Texas
  - Pfizer Investigational Site, Spring, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, West Jordan, Utah
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Bellevue, Washington
  - Pfizer Investigational Site, Puyallup, Washington
  - Pfizer Investigational Site, Tacoma, Washington